CLINICAL TRIAL: NCT03003195
Title: A Combined Phase I/II Study of a Carbohydrate Mimotope-Based Vaccine with MONTANIDE™ ISA 51 VG STERILE for Metastatic Cancer
Brief Title: The P10s-PADRE Basket Trial: Vaccination of Metastatic Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206265
Record Dates: First submitted 2016-12-19; First posted 2016-12-26 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2021-03

CONDITIONS: Neoplasms by Site; Metastatic Cancer
MeSH Terms: conditions — Neoplasms by Site; Neoplasm Metastasis | interventions — montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccination: P10s-PADRE/MONTANIDE ISA 51 VG (Experimental): 100mL vaccination on Weeks 1, 2, 3 and 8
  Interventions: Drug: P10s-PADRE

INTERVENTIONS:
Drug: P10s-PADRE — All research participants will receive the Mimotope P10s-PADRE/MONTANIDE ISA 51 VG vaccine via subcutaneous (SC) injection for a total of 4 vaccinations.
  Other Names: MONTANIDE ISA 51 VG

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of an investigational agent, P10s-PADRE, a peptide mimotope-based vaccine in subjects with metastatic cancer.

DETAILED DESCRIPTION:
After signing Institutional Review Board (IRB) approved consent, subjects with metastatic cancer will be enrolled. The vaccine doses will be prepared and dispensed by the University of Arkansas for Medical Sciences (UAMS) Pharmacy following the manufacturer's instructions. Subjects will receive 1.0 mL subcutaneous injections of the vaccine on 4 separate occasions. The vaccine will be administered at rotating sites on the limbs or abdomen. The study will last approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of all races with clinical Stage IV cancer of any type, staged according to American Joint Commission on Cancer (AJCC), sixth edition, receiving any line of standard treatment for the specific cancer and with stable disease or better for at least two months will be invited to participate.
* Subjects of all races with clinical Stage IV cancer of any type, staged according to American Joint Commission on Cancer (AJCC), sixth edition, who have no standard treatment options for the specific cancer (Patients whose standard of care consists of watchful waiting) and who fulfill the other eligibility criteria will be invited to participate.
* Measurable or evaluable disease.
* Patients with bone-only disease will be allowed to participate.
* Ages 18 years and older.
* ECOG Performance status 0, 1 or 2.
* White blood cells (WBC) count ≥ 3,000/mm3 within 3 weeks prior to registration
* Platelet count ≥ 100,000/mm3 prior to registration
* Serum glutamic-oxaloacetic transaminase (SGOT) ≤ 2 x institutional upper limit (IUL) of normal obtained within 3 weeks prior to registration or Aspartate aminotransferase test (AST) ≤ 2 x institutional upper limit (IUL) of normal obtained within 3 weeks prior to registration
* Bilirubin ≤ 2 x institutional upper limit (IUL) of normal obtained within 3 weeks prior to registration.
* Serum creatinine ≤ 1.8 mg/dl obtained within 3 weeks prior to registration.
* Must sign an informed consent document approved by UAMS Institutional Review Board (IRB).

Exclusion Criteria:

* Active infection requiring treatment with antibiotics.
* Existing diagnosis or history of organic brain syndrome that precludes participation in the full protocol.
* Existing diagnosis or history of significant impairment of basal cognitive function that might preclude participation in the full protocol.
* Other current malignancies. Subjects with prior history at any time of any in situ cancer, including lobular carcinoma in situ of the breast, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ, or basal or squamous skin cancer are eligible, provided they are disease-free of these other malignancies at the time of registration. Subjects with other malignancies - other than the one for which they are being treated - are eligible if they have been continuously disease free (from the old cancer) for ≥ 5 years prior to the time of registration.
* Existing diagnosis or history of autoimmune disorders or conditions of immunosuppression. This includes, but is not limited to, being treated with corticosteroids, including oral steroids (i.e. prednisone, dexamethasone [except when used as an antiemetic in standard therapy]), continuous use of topical steroid creams or ointments or any steroid-containing inhalers. Subjects who have been on systemic steroids will require a 6-week washout period. Subjects who discontinue the use of these classes of medication for at least 6 weeks prior to registration are eligible if, in the judgment of the treating physician, the subject is not likely to require these classes of drugs during the treatment period. Replacement doses of steroids for subjects with adrenal insufficiency are allowed.
* Pregnancy or breast feeding, due to the unknown effects of peptide/mimotope vaccines on a fetus or infant. Women of childbearing potential must have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study drug, and must be counseled to use an accepted and effective method of contraception while on treatment and for a period of 18 months after completing or discontinuing treatment. Accepted methods include oral contraceptives, barrier method, IUDs, and abstinence.
* Any other significant medical or psychiatric conditions which, in the opinion of the enrolling investigator, may interfere with consent or compliance of the treatment.
* Patients receiving checkpoint inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Immune Response | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Issam Makhoul, MD, Principal Investigator — University of Arkansas

IPD SHARING:
Plan to Share IPD: No